CLINICAL TRIAL: NCT03922893
Title: Discovery and Characterization of Susceptibility Genes in Adults and Children With Suspected Hereditary Cancer Predisposition
Brief Title: Discovering New Genetic Markers in Adults and Children Who May Be At Risk for Hereditary Forms of Cancer
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: New York Genome Center (Other)
Responsible Party: Sponsor
Other Study IDs: 19-133
Record Dates: First submitted 2019-04-18; First posted 2019-04-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Cancer
Keywords: Genetic evaluation; Germline genetic variant; Genetic cancer; Memorial Sloan Kettering Cancer Center; 19-133
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of biological specimens (DNA, RNA, tissue)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Proband: First individual in a family to consent to this protocol
  Interventions: Other: Family History Information; Genetic: ORAGENE; Genetic: Blood; Other: Skin Biopsy
- Family Member Participants: Family members of the proband will be approached to consent to this protocol
  Interventions: Other: Family History Information; Genetic: ORAGENE; Genetic: Blood; Other: Skin Biopsy

INTERVENTIONS:
Other: Family History Information — The family history ascertainment focuses on self-reported family history of first-, second-, and third-degree family members, including types of malignancies/ pre-malignant lesions and age at diagnosis.
Genetic: ORAGENE — Approximately 2-4mL of saliva may be collected in specialized Oragene DNA Self-Collection Kit tubes or buccal swab-based collection devices.
  Other Names: Saliva
Genetic: Blood — For select participants, 1-2 tubes of blood will be drawn for DNA and RNA analysis
Other: Skin Biopsy — In certain circumstances, for Memorial Sloan Kettering participants and their family members, it may be necessary to obtain a skin biopsy.

SUMMARY:
This study is being done to attempt to identify genetic mutations or other gene-based variations in adults and children who have cancer, or are likely to develop an inherited form of cancer, and potentially reduce their risk for cancer or treat the cancer earlier.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have undergone clinical and/or research genetic evaluation, found to have or not have a germline genetic variant (pathogenic, likely pathogenic, variant of uncertain/unknown significance, likely benign).
* Individuals with or without a personal history of malignant or pre-malignant lesions who demonstrate: a) clinical findings suggestive of a genetic cancer susceptibility syndrome including very early age at onset, multiple primary malignancies, or other features; and/or b) family histories suggestive of a genetic cancer susceptibility syndrome, or c) other features suggesting inherited etiology of malignancy as determined by the PI.
* Family members of the above participants. Both children (with parental consent as age appropriate) and adults are eligible to participation.
* Individuals may or may not be enrolled MSK patients; probands may be referred to (or self-referred to) the study and may be enrolled at discretion of the PI and if able to provide informed consent.
* Biospecimens derived from deceased family members may be used for research in this study if consent if provided by the executor of the estate of that individual.

Exclusion Criteria:

* Patients will be excluded from this study if he/she has physical, cognitive or psychiatric conditions that interfere with ability to give meaningful informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants will be identified by members of the Clinical Genetics Service from the following sources: a) MSK patients previously tested through MSK IMPACT #12-245 protocol; b) MSK patients referred to the Clinical Genetics Service by an MSK physician, outside physician, or self-referral; c) non-MSKCC patients referred or self-referred to the Clinical Genetics Service or directly to the P.I. and identified as candidates for participation in this study; d) family members of probands identified by the study team to be informative for research purposed.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2019-04-17 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Discovery of novel cancer susceptibility genes | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Offit, MD, MPH, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org